CLINICAL TRIAL: NCT07009548
Title: CytoGam® as Adjuvant Therapy to Prevent or Attenuate Human Cytomegalovirus (CMV) Infection and Disease in Solid Organ Transplant Recipients
Brief Title: CytoGam for CMV Infection or Disease in Solid Organ Transplant Recipients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Fernanda P Silveira, MD, MS (Other)
Collaborators: Kamada, Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Fernanda P Silveira, MD, MS, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25030118
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Cytomegalovirus (CMV) Infection
Keywords: cytomegalovirus; CMV; CytoGam; immunoglobulin; organ transplant
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — cytomegalovirus-specific hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CytoGam for primary CMV infection after lung or liver transplantation or for high viral load (Experimental): There are 3 cohorts in this treatment arm:
  * CMV D+/R- lung transplant recipients who develop any level of CMV DNAemia after discontinuation of valganciclovir prophylaxis and who have not yet received antiviral treatment for greater than 14 days will receive one dose of CytoGam.
  * CMV D+/R- liver transplant recipients on pre-emptive therapy who develop any level of detectable CMV DNAemia and who have not yet received antiviral treatment for greater than 14 days will receive one dose of CytoGam.
  * Recipients of any solid organ transplant who have CMV DNAemia ≥ 50,000 IU/ml, with or without CMV disease, and who have not yet received antiviral therapy for greater than 14 days will receive one dose of CytoGam.
  For all cohorts the choice and duration of antiviral therapy will be at the discretion of the treating physician.
  Interventions: Drug: Cytogam

INTERVENTIONS:
Drug: Cytogam — CytoGam 150 mg/kg intravenously (IV) administered as a single dose
  Other Names: Cytomegalovirus Immune Globulin Intravenous; CMV-IGIV

SUMMARY:
Cytomegalovirus (CMV) is a significant opportunistic pathogen and a major cause of morbidity and mortality in solid organ transplant recipients. CytoGam - Cytomegalovirus Immune Globulin Intravenous (CMV-IGIV), is an immunoglobulin G containing a standardized amount of antibody against CMV. CytoGam is obtained from pooled adult human plasma that has been selected for high anti-CMV titers. This study will evaluate if administration of CytoGam to organ transplant recipients with CMV infection, along with standard of care antiviral medication, leads to faster clearance of CMV from the blood, prevents the development of antiviral resistance, and decreases the rate of recurrence of CMV infection.

DETAILED DESCRIPTION:
Interventional, open-label, single center, pilot study to test the effect of CytoGam on CMV viremia clearance in organ transplant recipients with high CMV viral load and in CMV D+/R- lung and liver transplant recipients with primary CMV infection.

CMV D+/R- lung transplant recipients who develop any level of CMV DNAemia after discontinuation of valganciclovir prophylaxis and who have not yet received antiviral treatment for greater than 14 days will receive one dose of CytoGam. The choice and duration of antiviral therapy will be at the discretion of the treating physician. Patients will be followed until 2 weekly negative CMV PCRs, discontinuation of antiviral, or 1 year from CytoGam infusion, whichever is longer.

CMV D+/R- liver transplant recipients on pre-emptive therapy who develop any level of detectable CMV DNAemia and who have not yet received antiviral treatment for greater than 14 days will receive one dose of CytoGam. The choice and duration of antiviral therapy will be at the discretion of the treating physician. Patients will be followed until 2 weekly negative CMV PCRs, discontinuation of antiviral, or 1 year from CytoGam infusion, whichever is longer.

Recipients of any solid organ transplant who have CMV DNAemia ≥ 50,000 IU/ml, with or without CMV disease, and who have not yet received antiviral therapy for greater than 14 days will receive one dose of CytoGam. The choice and duration of antiviral therapy will be at the discretion of the treating physician. Patients will be followed until 2 weekly negative CMV PCRs, discontinuation of antiviral, or 1 year from CytoGam infusion, whichever is longer.

ELIGIBILITY:
Inclusion Criteria - all study arms:

* Written informed consent obtained from the subject before any trial-related procedures are performed
* >= 18 years and <= 75 years of age at time of consent
* Able to perform routine blood testing (standard care for transplant recipients)
* Understands and can read English

Inclusion criteria - high viral load arm:

* Recipient of an organ transplant (lung, heart, liver, kidney, pancreas, intestine alone or in combination) and on immunosuppression
* CMV DNAemia ≥ 50,000 IU/ml in the first 2 weeks of CMV antiviral treatment with CMV antiviral dose appropriately adjusted for renal function

Inclusion criteria - CMV primary infection after liver transplantation arm:

- Liver transplant recipients who are CMV IgG negative and received a CMV IgG positive donor (CMV D+/R-) with a primary CMV infection, defined as detected CMV DNAemia, including detected but below the limit of quantitation

Inclusion criteria - CMV primary infection after lung transplantation arm:

- Lung transplant recipients who are CMV D+/R- with a primary CMV infection after discontinuation of CMV antiviral prophylaxis, defined as detected CMV DNAemia, including detected but below the limit of quantitation

Exclusion Criteria:

* History of hypersensitivity to or a prior severe reaction associated with the administration of CytoGam or other human immunoglobulin preparation
* Receipt of effective CMV antiviral treatment, appropriately adjusted for renal function, for greater than or equal to 14 days prior to enrollment
* Selective IgA deficiency, as they may produce antibodies against immunoglobulin A (IgA), leading to potential anaphylactic reactions upon administration of blood products containing IgA, including CMV immunoglobulin (e.g. CytoGam or similar)
* Prior history of hematopoietic cell transplant
* Pregnancy
* Participation in another interventional clinical trial at time of consent or within 30 days prior to study consent
* Any condition which, in the judgement of the investigator, would make administration of CytoGam unsafe

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Time to CMV DNAemia clearance | 1 year
  Time from administration of CytoGam to CMV DNAemia clearance, defined as CMV PCR not detected or detected but below the limit of quantitation

SECONDARY OUTCOMES:
Duration of antiviral therapy | 1 year
  Duration of administration of antiviral therapy
Number of participants with de novo ganciclovir-resistance | 1 year
  Participants who develop laboratory-confirmed ganciclovir-resistance after CytoGam administration
CMV recurrence | Within 90 days of administration of CytoGam
  Recurrence of and time to CMV DNAemia greater than the lower limit of quantification

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Silveira, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data outside of our investigative team and collaborators. Aggregate data will be shared in publications as appropriate.